CLINICAL TRIAL: NCT06914453
Title: A Comparative Study of Air-Q3 and Ambu AuraGain Supraglottic Airway Device in Patients Undergoing Elective Surgery Under General Anaesthesia: A Randomised Controlled Trial
Brief Title: A Randomised Controlled Trial to Compare Two Supraglottic Airway Devices (Ambu AuraGain vs Air Q-3) in Terms of Performance Characteristics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Lee Shu Ren, Medical Doctor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UMalaya (MREC 2024426-13665)
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Oropharyngeal Leak Pressure; Supraglottic Airway; Elective Surgery; General Anaesthesia
Keywords: Ambu AuraGain; Supraglottic Airway Device; General Anaesthesia; Oropharyngeal leak pressure; Laryngeal Alignment; Air-Q3

STUDY DESIGN:
Intervention Model Description: Two Types of Supraglottic Airway Devices (Ambu AuraGain and Air Q-3) are involved. A total of 90 patients will be randomised using a computer-generated randomisation table to either receive Air-Q3 or Ambu AuraGain. 45 patients in each group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambu AuraGain (Active Comparator): Patients in this group, once under general anaesthesia, will have this supraglottic airway device inserted to maintain airway patency and maintenance of general anaesthesia.
  Interventions: Device: Ambu AuraGain Supraglottic Airway Device
- Air Q-3 (Active Comparator): Patients in this group, once under general anaesthesia, will have this supraglottic airway device inserted to maintain airway patency and maintenance of general anaesthesia.
  Interventions: Device: Air Q-3 Supraglottic Airway Device

INTERVENTIONS:
Device: Air Q-3 Supraglottic Airway Device — Oropharyngeal leak pressure and other performance characteristics including time to insertion, first-pass success rate, ease of orogastric tube (OGT) insertion, laryngeal alignment using a fiberoptic scope, and incidence of postoperative sore throat.
  Arms: Air Q-3
Device: Ambu AuraGain Supraglottic Airway Device — Oropharyngeal Leak Pressure and other performance characteristics including time to insertion, first-pass success rate, ease of orogastric tube (OGT) insertion, laryngeal alignment using a fiberoptic scope, and incidence of postoperative sore throat.
  Arms: Ambu AuraGain

SUMMARY:
A supraglottic airway device (SAD) functions as a temporary device to maintain the patency of airway during the administration of anaesthesia. The Ambu AuraGain (Ambu, Ballerup, Denmark) is a second generation SAD, since introduced in 2014, has been widely used in clinical practice. The Ambu AuraGain is an anatomically curved, single-use supraglottic airway device that features a port for orogastric tube insertion and it is a conduit for intubation as well. It is also associated with fast insertion times and high seal pressures. The Air-Q3, on the other hand, is relatively new SAD, however rather similar to Ambu AuraGain, it is also anatomically curved with a built-up mask heel for improved seal and it serves as a conduit for intubation as it features a unique endotracheal tube ramp and epiglottis elevator which aids in fast easy and safe intubation. It also features a port for orogastric tube insertion. Given the relatively recent introduction of the Air-Q3 into the market, there exists a paucity of comprehensive data regarding its efficacy. Meanwhile, the Ambu AuraGain stands as one of the most frequently utilised SAD, especially in our centre. This randomized controlled trial aims to compare the performance characteristics of the Ambu AuraGain and Air Q-3 in 90 patients undergoing surgery under general anaesthesia. The primary objective is to evaluate oropharyngeal leak pressure (OLP), while secondary objectives includes time to insertion, first-pass success rate, ease of orogastric tube (OGT) insertion, laryngeal alignment using a fiberoptic scope, and incidence of postoperative complications.

DETAILED DESCRIPTION:
Preoperative assessment, encompassing history taking, physical examination, laboratory investigation, and a comprehensive explanation of the study, will be conducted the day prior to surgery. Patients will be instructed to fast for 6 hours for solid foods and 2 hours for clear fluids before elective surgery.

Patients will be randomly allocated to either the Air-Q3 group (n = 45) or the Ambu AuraGain group (n = 45) using a computer-generated randomization table. After recruitment, the enrolling investigator opens the sealed opaque envelopes that concealed group allocation. Patients will be blinded to their group allocation. Patients will not receive any premedication and will be positioned supine on the operating table, head in neutral position, rested on a gel head ring. Standard monitoring including basic physiological variables, including electrocardiography, pulse oximetry, non-invasive blood pressure monitoring, and end-tidal oxygen measurement using a circle circuit ventilator (Datex Ohmeda, Aespire, Marquet), will be performed prior to anaesthesia induction.

Following establishment of intravenous access, a standard anaesthesia induction protocol will be followed, involving preoxygenation with 100% inspired oxygen for 3 minutes, intravenous administration of Fentanyl (1-2mcg/kg), and Propofol (2-3mg/kg) until loss of consciousness. Subsequently, either the Air-Q3 or Ambu AuraGain will be lubricated and prepared according to manufacturers' recommendations. The airway device will be inserted when the jaw is sufficiently relaxed. The cuff of each device will be inflated with air to a final cuff pressure of 60cmH20. The cuff pressure is measured by a handheld manometer, The airway device insertions will be performed by experienced staff anaesthesiologists with more than ten years experience with supraglottic airway management, who had performed at least 10 Air-Q3 insertions prior to trial commencement.

SAD size selection will adhere to manufacturers' recommendations based on the patient's ideal body weight. Insertion time will be recorded from facemask removal until the presence of square wave capnography tracing. The presence of square wave capnography tracing denotes successful establishment of effective ventilation. Otherwise, the device will be removed completely for another insertion attempt. Failure to insert the SAD after two attempts will be deemed a failure.

After successful insertion of the airway device, it will be secured with tape over the patient's check. A gel plug is applied to the orogastric port and a suprasternal notch test (gentle tapping over the suprasternal notch results in the gel to pulsate, confirming tip location behind the cricoid cartilage) will be done to confirm placement. A 14 French gauge gastric tube, pre lubricated with a water soluble lubricant will be inserted through the nasogastric port for both devices. The ease of insertion will be graded from 1 to 3 (1 = easy, 2 = difficult, 3 = impossible). After successful insertion of the airway device, it will be secured with tape over the patient's check. A gel plug is applied to the orogastric port and a suprasternal notch test (gentle tapping over the suprasternal notch results in the gel to pulsate, confirming tip location behind the cricoid cartilage) will be done to confirm placement. A 14 French gauge gastric tube, pre lubricated with a water soluble lubricant will be inserted through the nasogastric port for both devices. The ease of insertion will be graded from 1 to 3 (1 = easy, 2 = difficult, 3 = impossible). Confirmation of correct orogastric tube placement will be established through aspiration of gastric contents or epigastric auscultation.

Oropharyngeal leak pressure will be determined by transiently halting ventilation and closing the adjustable pressure limiting valve up to 30cmH2O with a fresh gas flow of 3L/min. The airway pressure at equilibrium or when audible air leak is heard from the throat is recorded.

Following successful SAD insertion, fibreoptic scope assessment will be conducted to evaluate LMA placement, graded based on the standardized scale by Brimacombe:

1. Vocal cords not seen
2. Vocal cords plus anterior epiglottis visible
3. Vocal cords plus posterior epiglottis visible
4. Only vocal cords visible Maintenance of general anaesthesia will be with sevoflurane with minimum alveolar concentration 1 - 2 in an oxygen-air mixture.

Postoperatively, patients will be monitored in the recovery room, with physiological variables including non-invasive blood pressure, heart rate, pulse oximetry, and respiratory rate continuously monitored. Upon full consciousness and recovery, a blinded investigator will assess for the presence of sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 to 65 years) of either sex, who are scheduled for an elective surgery under general anaesthesia
* Patients with ASA physical status of I or II.

Exclusion Criteria:

* Patients with anticipated difficult airway (Airway Difficulty Score >8)
* Patients with high risk of aspiration and regurgitation
* Patients with body mass index (BMI) > 40kg/m2
* Patients who exhibit evidence of upper respiratory tract infection
* Patients with history of radiotherapy to the neck
* Patients who are pregnant
* Patients who are unable or unwilling to consent for the study
* Patients who are mentally challenged and unable to understand the study instructions
* Planned operating time more than 4 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) of the Air-Q3 and Ambu AuraGain supraglottic airway device | After induction of general anaesthesia until successful insertion of supraglottic airway device
  After induction of general anaesthesia, either one supraglottic airway device will be inserted, Oropharyngeal leak pressure will be determined by transiently halting ventilation and closing the adjustable pressure limiting valve up to 30cmH2O with a fresh gas flow of 3L/min. The airway pressure at equilibrium or when audible air leak is heard from the throat is recorded.

SECONDARY OUTCOMES:
Other performance characteristics in terms of time to insertion, first pass success rate, ease of orogastric tube (OGT) insertion. | After induction of anaesthesia until comfirmation of correct orogastric tube placement will be established through aspiration of gastric contents or epigastric auscultation
  Time of insertion will be recorded during the insertion of the airway device, the number of attempts to successful insertion will also be recorded. The ease of insertion of gastric tube will be graded from 1 to 3 (1 = easy, 2 = difficult, 3 = impossible).
Laryngeal alignment using fibreoptic scope by employing the standardised scale developed by Brimacombe | After insertion of supraglottic airway device till performing fibreoptic scope assessment
  Following successful SAD insertion, fibreoptic scope assessment will be conducted to evaluate LMA placement, graded based on the standardized scale by Brimacombe:
  1. Vocal cords not seen
  2. Vocal cords plus anterior epiglottis visible
  3. Vocal cords plus posterior epiglottis visible
  4. Only vocal cords visible
Incidence of complications of using both SADs such as post operative sore throat | From extubation until full consciousness in recovery area
  Post extubation, patient will be assessed for presence of sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Ina Ismiarti Shariffuddin, Clinical Professor, Study Director — Univerisity Malaya
Locations (1):
- Department of Anaesthesiology, Faculty of Medicine, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta R, Mahajan R, Jatinder M, Gulati S, Mehta A, Nazir R. A comparison between ProSeal laryngeal mask airway and Air-Q Blocker in patients undergoing elective laparoscopic cholecystectomy. J Anaesthesiol Clin Pharmacol. 2019 Jul-Sep;35(3):340-347. doi: 10.4103/joacp.JOACP_397_17. PMID 31543582
- [Background] Preece G, Ng I, Lee K, Mezzavia P, Krieser R, Williams DL, Stewart O, Segal R. A randomised controlled trial comparing fibreoptic-guided tracheal intubation through two supraglottic devices: Ambu(R) AuraGain laryngeal mask and LMA(R) Fastrach. Anaesth Intensive Care. 2018 Sep;46(5):474-479. doi: 10.1177/0310057X1804600508. PMID 30189821
- [Background] Singh A, Bhalotra AR, Anand R. A comparative evaluation of ProSeal laryngeal mask airway, I-gel and Supreme laryngeal mask airway in adult patients undergoing elective surgery: A randomised trial. Indian J Anaesth. 2018 Nov;62(11):858-864. doi: 10.4103/ija.IJA_153_18. PMID 30532321
- [Background] Shariffuddin II, Teoh WH, Tang E, Hashim N, Loh PS. Ambu(R) AuraGain versus LMA Supreme Second Seal: a randomised controlled trial comparing oropharyngeal leak pressures and gastric drain functionality in spontaneously breathing patients. Anaesth Intensive Care. 2017 Mar;45(2):244-250. doi: 10.1177/0310057X1704500215. PMID 28267947
- [Background] Che Omar S, Hardy Mohamad Zaini R, Fui Wong T, Nazaruddin W Hassan WM. Comparison of the Air-Q intubating laryngeal mask airway and the Ambu AuraGain laryngeal mask airway as a conduit for fibreoptic assisted endotracheal intubation for simulated cervical spine injury. Anaesthesiol Intensive Ther. 2021;53(3):241-245. doi: 10.5114/ait.2021.105759. PMID 34006053
- [Background] Jindal S, Mittal A, Anand LK, Singh M, Kapoor D. Comparative evaluation of Air-Q blocker and Proseal laryngeal mask airway in patients undergoing elective surgery under general anaesthesia: A randomised controlled trial. Indian J Anaesth. 2021 Mar;65(Suppl 1):S20-S26. doi: 10.4103/ija.IJA_1254_20. Epub 2021 Mar 20. PMID 33814586
- [Background] Brimacombe J, Berry A. A proposed fiber-optic scoring system to standardize the assessment of laryngeal mask airway position. Anesth Analg. 1993 Feb;76(2):457. No abstract available. PMID 8424538
- See also: Ambu AuraGain Official Website — https://www.ambu.com/airway-management-and-anaesthesia/laryngeal-masks/product/ambu-auragain-disposable-laryngeal-mask
- See also: Air Q-3 Official Website — https://www.myairlife.com/product/air-q3-intubating-laryngeal-airway